CLINICAL TRIAL: NCT02726750
Title: Observational Prospective Research Study In Monoclonal Gammopathies leadINg to Myeloma (ORIGIN Study)
Brief Title: Observational Prospective Research Study In Monoclonal Gammopathies leadINg to Myeloma
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA15-0575; NCI-2020-07336 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA15-0575 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection): Patients undergo collection of blood samples every 6 months for 3 years. Patients may also undergo a biopsy, x-rays, PET/CT scans, and/or MRI scans to check the status of disease at the discretion of the treating physician.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
The goal of this study is to find markers that may help to predict why some patients who have monoclonal gammopathy of unknown significance (MGUS) or smoldering multiple myeloma (SMM) that have no signs or symptoms of disease (asymptomatic) develop multiple myeloma, while others do not. Studying markers such as age, level of proteins in blood, percent of abnormal blood cells in the bone marrow, genes in the abnormal blood cells, and bone abnormalities may help researchers to validate clinical and genomic predictors for future use in clinical practice.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of progression to multiple myeloma after 3 years of follow up.

SECONDARY OBJECTIVES:

I. To describe baseline patient characteristics and clinical variables. II. To identify molecular and genetic correlates that may predict for progression to multiple myeloma (MM).

OUTLINE:

Patients undergo collection of blood samples every 6 months for 3 years. Patients may also undergo a biopsy, x-rays, positron emission tomography (PET)/computed tomography (CT) scans, and/or magnetic resonance imaging (MRI) scans to check the status of disease at the discretion of the treating physician.

After completion of 3 years on study, patients are followed up every 6-12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with monoclonal gammopathy of unknown significance. Both criteria must be met:

  * Serum monoclonal protein < 3 g/dL or urinary monoclonal protein < 500 mg per 24 hours and clonal bone marrow plasma cells < 10%
  * Absence of myeloma defining events or amyloidosis
* Patients with smoldering multiple myeloma. Both criteria must be met:

  * Serum monoclonal protein >= 3 g/dL or urinary monoclonal protein >= 500 mg per 24 hours and/or clonal bone marrow plasma cells 10-60%
  * Absence of myeloma defining events or amyloidosis

Exclusion Criteria:

* Evidence of myeloma defining events or biomarkers of malignancy due to underlying plasma cell proliferative disorder meeting at least one of the following

  * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  * Renal Insufficiency: creatinine clearance < 40 ml/min or serum creatinine > 2 mg/dL
  * Anemia: hemoglobin value < 10 g/dL or 2 g/dL < normal reference
  * Bone lesions: one or more osteolytic lesions on skeletal radiography, computerized tomography (CT) or 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography CT (PET-CT)
  * Clonal bone marrow plasma cell percentage >= 60%
  * Involved:uninvolved serum free light chain ratio >= 100 measured by Freelite assay (The Binding Site Group, Birmingham, United Kingdom [UK])
  * > 1 focal lesions on magnetic resonance imaging (MRI) studies (each focal lesion must be 5 mm or more in size)
* Prior or concurrent systemic treatment for asymptomatic monoclonal gammopathies

  * Bisphosphonates are permitted
  * Radiotherapy is not permitted
  * Prior treatment with chemotherapy or investigational agents for asymptomatic gammopathies is not permitted
* Plasma cell leukemia
* Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with monoclonal gammopathy of unknown significance and/or smoldering multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-12-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of progression to multiple myeloma (MM) | 3 years
  Kaplan-Meier method will be used to estimate time to MM progression. Log-rank test will be used to evaluate the difference in rate of progression between/among patient groups.
Progression free survival | 3 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be used to evaluate the difference in rate of progression free survival between/among patient groups.
Overall survival | 3 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be used to evaluate the difference in rate of overall survival between/among patient groups.

SECONDARY OUTCOMES:
Baseline patient characteristics and clinical variables | Baseline
  Summary statistics including mean, standard deviation, median, and range will be provided for continuous variables. Frequency counts and percentages will be used to summarize categorical variables.
Molecular and genetic profile analysis | 3 years
  Will study the correlation of molecular and genetic profiles with time to MM progression.

OTHER OUTCOMES:
Molecular profiling analysis of patients who develop MM | 3 years
  Analysis will include whole exome sequencing and gene expression profiling and cellular (including flow cytometry) profiling using bone marrow and peripheral blood samples.
Immune characterization of patients who develop MM | 3 years
  Analysis will include cell surface and functional studies of dendritic, T-, B-, natural killer (NK)- and NKT-cells using peripheral blood samples.
Immune characterization of patients who develop MM | 3 years
  Analysis will include cell surface and functional studies of dendritic, T-, B-, NK- and NKT-cells using bone marrow samples.

CONTACTS AND LOCATIONS:
Overall Officials: Krin Patel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org